CLINICAL TRIAL: NCT01129895
Title: Promoting Health by Self Experience (PHASE) Randomized Controlled Trial
Acronym: PHASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unilever Israel (Industry)
Responsible Party: Danit R Shahar, Ben-Gurion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: unilever-0410-OL
Record Dates: First submitted 2010-05-22; First posted 2010-05-25 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Personal Experience and Personal Initiation Program; Health Prevention Activities; Impact on Patients
MeSH Terms: interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health promotion (Experimental): 5 workshops on the initiation of health prevention projects in each clinic will be organized by the intervention team and than the clinic will be followed by the intervention team for 6 months.
  Interventions: Behavioral: Health promotion
- Promoting Health (No Intervention): No intervention follow-up only

INTERVENTIONS:
Behavioral: Health promotion — In each intervention clinic 5 workshops on the initiation of health prevention projects in each clinic will be organized by the intervention team and than the clinic will be followed by the intervention team for 6 months.
  Arms: Health promotion

SUMMARY:
Promoting Health by Self Experience (PHASE) randomized controlled trial

Study Hypothesis:

A personal experience in health promotion will affect the health prevention activities of the health providers and thus will impact their prevention activities toward their patients compared with a control (no-intervention) group.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of a personal experience and personal initiation program on the health prevention activities of the health providers and the following impact on their patients compared with a control (no-intervention) group.

Methods: A randomized controlled trial Randomization: Health providers of all disciplines will be recruited from 10 clinics of Clalit Health Services, Dan district and randomized using cluster (by clinic) randomization, into an intervention and a control group. In each clinic 15 health care providers and 50 patients will be interviewed providing a total of 150 health care providers and 500 patients.

Intervention: The intervention will be delivered by psychologists and social workers trained in group facilitation and experimental learning. The program is based on theories of experimental learning and Bridges model of change. In each intervention clinic 5 workshops on the initiation of health prevention projects in each clinic will be organized by the intervention team and than the clinic will be followed by the intervention team for 6 months. No intervention will be provided to the control clinics.

Outcomes: changes in quality measurements of both intervention and non-intervention clinics. Among health providers changes in attitudes, personal views and life style as well as health prevention activities will be assessed by questionnaires. A random sample of 50 patients age 21-50 from each of the participating clinics will be selected and interviewed using a questionnaire. The questionnaires will include questions regarding the administration of screening tests, treatment of abnormal measurements, life style changes and satisfaction with the performance of the clinic and health care providers. The evaluation for both health care providers and patients will be performed at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Health providers in selected clinics
* Patients age 21-50 in selected clinics

Exclusion Criteria:

* Patients age younger than 21 and older than 50
* Health providers from clinics not in the area of the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 650 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Promoting Health randomized controlled trial | 6 months
  Changes in quality measurements Changes in attitudes, personal views and life style as well as health prevention activities

CONTACTS AND LOCATIONS:
Overall Officials: Iris Shai, PhD, Principal Investigator — Ben-Gurion University of the Negev; Danit R Shahar, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Clalit Health Services, Petah Tikva, Israel, Israel

REFERENCES:
- [Derived] Shai I, Erlich D, Cohen AD, Urbach M, Yosef N, Levy O, Shahar DR. The effect of personal lifestyle intervention among health care providers on their patients and clinics; the Promoting Health by Self Experience (PHASE) randomized controlled intervention trial. Prev Med. 2012 Oct;55(4):285-291. doi: 10.1016/j.ypmed.2012.08.001. Epub 2012 Aug 12. PMID 22906808